CLINICAL TRIAL: NCT03784248
Title: Mediterranean Visceral Leishmaniasis With Leishmania Infantum: Genetic Characterization of the Host Parasite in Relation to Asymptomatic Human Carriage
Brief Title: Mediterranean Visceral Leishmaniasis With Leishmania Infantum
Acronym: AsymptoGen
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 17-API-02
Record Dates: First submitted 2018-11-20; First posted 2018-12-21 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Leishmaniasis
MeSH Terms: conditions — Leishmaniasis | interventions — Blood Donation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- asymptomatic carrier
  Interventions: Other: blood donation and isolation of leuco-platelet layers
- uninfected subjects
  Interventions: Other: blood donation and isolation of leuco-platelet layers

INTERVENTIONS:
Other: blood donation and isolation of leuco-platelet layers — patients donating blood. Blood bags will be treated and leuco-platelet coatings will be sent to Nice

SUMMARY:
L. infantum leishmaniasis is endemic in the South of France. For several years, there has been an expansion of the territory of sandflies (vector of leishmaniasis), with the appearance of cases of canine leishmaniasis in new outbreaks: West of the Occitania region (South-West). The transition from asymptomatic to disease depends largely on the immune status of the carrier, but many other factors specific to the parasite and host remain poorly defined. Asymptomatic carriage is present in a large majority of infected subjects, however, to date, only parasite isolates causing the patent form have been characterized.

In this PHRC, the team wishes to study the genetics of parasite isolates present in asymptomatic carriers of the Alpes-Maritimes outbreak and the new Occitanie outbreak as well as the genetics of the host.

The primary objective is the genetic characterization of L. infantum isolates by the microsatellite method, present in asymptomatic carriers in southeast and southwestern France.

The secondary objectives are:

1. Comparison of the genetic profiles of L. infantum isolates, by microsatellite method, from asymptomatic carriers of the new Southwestern outbreak with isolates from asymptomatic carriers of the historical Southwestern outbreak.
2. Comparison of the genetic profiles of L. infantum isolates, by the microsatellite method, present in asymptomatic carriers in the Southeast with the profiles of isolates present in patients in the same outbreak, for whom a microsatellite study has already been obtained previously.
3. the team is also conducting a preliminary study of the host genetic factors that would be associated with asymptomatic carriage by studying the association between potential host-related genetic risk factors (HLA typing, NLRP3 gene study) and asymptomatic carriage. Indeed, a recent study showed that the NLRP3 gene prevents the development of the patent form of leishmaniasis in the mouse model. This preliminary genetic study will identify potential host-related factors associated with asymptomatic carriage.

To meet these objectives, leuco-platelet layer parasites (CLP) obtained via EFS from the 2 sources of interest will be isolated.

This project is a research not involving the human person. It is multicentric and non-randomized.

As a result of this research, isolates from asymptomatic carriers of the historical outbreak will be studied and compared to those present in new endemic outbreaks, as well as to those of patients already studied in a previous study. A better knowledge of parasites circulating in asymptomatic carriers will make it possible to study in a comprehensive way the risk factors associated with the parasite. In addition, the study of asymptomatic carrying in new endemic outbreaks such as Occitania is very original, since no human studies have yet been undertaken in this region. The results obtained in this PHRC will be used to understand the factors associated with the development of visceral leishmaniasis.

ELIGIBILITY:
Inclusion Criteria:

* Meet EFS blood donation criteria
* Provenance:

Department of Alpes-Maritimes, Var and Bouches du Rhône, for the historical endemic outbreak Department of Gers, Tarn-et-Garonne and Lot for the new Occitanie household

- Donor who has signed genetic consent

Exclusion Criteria:

* criteria for EFS blood donation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anyone aged 18 to 70, who weighs more than 50 kg and is recognized as fit following the predon interview, can donate blood.
  Men can give up to 6 times a year and women up to 4 times. Between two blood donations, a minimum of 8 weeks must be respected.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
genetic level characterization of the isolates of L. infantum | 6 months
  To characterize at the genetic level the isolates of L. infantum present in asymptomatic carriers in South-East and South-West France, it will be studied12 microsatellite loci by PCR - laboratory tests

CONTACTS AND LOCATIONS:
Locations (1):
- Nice Hospital, Nice, France